CLINICAL TRIAL: NCT05396976
Title: The Effect of Yoga and Progressive Muscle Relaxation Exercise Practices on Menstrual Symptoms, Depression, Anxiety and Stress in University Students: A Randomized Controlled Trial
Brief Title: The Effect of Yoga and Progressive Muscle Relaxation Exercise Practices on Premenstrual Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Arzu Abiç, Asist. Prof. Dr, Eastern Mediterranean University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: ETK00-2022-0100
Record Dates: First submitted 2022-04-28; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Syndrome; Yoga; Muscle Relaxation Exercise Practices; Depression, anxiety and stress
MeSH Terms: conditions — Premenstrual Syndrome; Depression; Anxiety Disorders | interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Yoga Group (Experimental): Yoga practice will be done two days a week for 10 weeks.
  Interventions: Behavioral: Yoga and Muscle Relaxation Exercise Practices
- control group (No Intervention): no intervention
- Muscle Relaxation Exercise Practices Group (Experimental): Muscle Relaxation Exercise Practices will be done two days a week for 10 weeks.
  Interventions: Behavioral: Yoga and Muscle Relaxation Exercise Practices
- Yoga and Muscle Relaxation Exercise Practices Group (Experimental): Yoga and Muscle Relaxation Exercise Practices will be done two days a week for 10 weeks.
  Interventions: Behavioral: Yoga and Muscle Relaxation Exercise Practices

INTERVENTIONS:
Behavioral: Yoga and Muscle Relaxation Exercise Practices — Yoga and Muscle Relaxation Exercise Practices will be done two days a week for 10 weeks.
  Arms: Muscle Relaxation Exercise Practices Group; Yoga Group; Yoga and Muscle Relaxation Exercise Practices Group

SUMMARY:
Yoga and progressive relaxation exercises are seen as a valuable approach for the management of PMS, which is very common in young women and has significant negative effects on academic participation, social activities and quality of life. Despite the conclusion that yoga and progressive relaxation exercises are an effective method in the treatment of PMS in a significant part of the studies in the literature, it is mentioned that the data are insufficient in terms of method and methodology and the necessity of studies that can support the results. In this study, it was aimed to determine the effects of yoga and progressive muscle relaxation exercises on menstrual symptoms, depression, anxiety and stress in university students with premenstrual syndrome.

DETAILED DESCRIPTION:
Menstrual cycle is defined as hormonal and physical changes that continue from menarche to menopause, affecting the whole organism, especially the reproductive organs. During this period, which is necessary for the normal continuation of female reproductive functions and occurs periodically every month, women encounter many menstrual problems. Premenstrual syndrome (PMS), one of the most common problems, is defined as the changes that are associated with the luteal phase of the menstrual cycle and that affect a woman's life in a regular and cyclical way, physically, emotionally and behaviorally.It is stated that PMS, which is very common in the society, affects close family relations, social life, work performance and work relations. The most common symptoms are; muscle, stomach and headache, breast tenderness, weight gain, intense desire for certain foods, appetite change, acne, edema, fatigue, mood swings, emotionality, irritability. It is known that the mental health of women who are physiologically affected by PMS will also be affected by the syndrome and bring along mental problems. Schmelzer stated in his study that the emergence of depressive thoughts and emotions in the premenstrual period is one of the most common PMS symptoms. In many studies examining the relationship between mental health and PMS, it has been found that there is a positive and significant relationship between PMS and depression level. One of these studies, Uran et al., in a study conducted with 55 people with an average age of 15, stated that the most common psychological factors accompanying PMS were irritability and anger level. As can be seen, PMS has negative effects on both mental health and physical health. Although many areas of women with PMS are negatively affected in their daily lives and its incidence is high, very few of them receive professional help and medical care. At the same time, their quality of life is also declining. It is known that women often resort to non-pharmacological methods instead of receiving professional health care, since PMS is considered to be a physiologically normal condition with a traditional point of view.In addition, undesirable effects of medical treatments in coping with PMS are not preferred by women because they bring many health risks. Women can use many non-invasive and risk-free integrated treatment methods (such as heat treatments, exercise, aromatherapy, phytotherapy, Transcutaneous Electrical Nerve Stimulation, acupuncture, acupressure, yoga, progressive relaxation exercises, massage, relaxation techniques, reflexology, reiki) in coping with PMS. ) are more oriented. One of these methods, yoga, is a practice that includes deep breathing, meditation, stretching exercises and posture poses based on the unity of mind and body. It is emphasized that yoga exercises reverse the negative effects of stress on the immune system, improve inflammatory processes, reduce symptoms such as pain and insomnia, and improve quality of life, thanks to the balance, stretching, relaxation and strengthening components.In Yang and Kim's study with undergraduate nursing students with primary dysmenorrhea, a 60-minute yoga program was applied once a week for 12 weeks. As a result of the study, it was determined that menstrual pain decreased significantly in the intervention group compared to the control group. Yonglitthipagon et al. found that yoga exercise applied to women with primary dysmenorrhea between the ages of 18-22 for 30 minutes twice a week for 12 weeks reduced menstrual pain and increased physical fitness and quality of life. It has also been reported in studies that progressive relaxation exercises have a reducing effect on depression, stress and anxiety. Yoga and progressive relaxation exercises are seen as a valuable approach for the management of PMS, which is very common in young women and has significant negative effects on academic participation, social activities and quality of life. Although it is concluded that yoga and progressive relaxation exercises are an effective method in the treatment of PMS in a significant part of the studies in the literature, it is mentioned that the data are insufficient in terms of method and methodology and the necessity of studies that can support the results. In this study, it was aimed to determine the effects of yoga and progressive muscle relaxation exercises on menstrual symptoms, depression, anxiety and stress in university students with premenstrual syndrome.

ELIGIBILITY:
Inclusion Criteria:

Filling the data collection tools and not having an obstacle that would cause communication difficulties in the interviews Having a score of 110 or more from the PMS scale in the data collection form Voluntary consent to participate in the study Having a regular menstrual period (occurring at intervals of 21-35 days and lasting 3-8 days), Being a second and third year nursing student be over 18 years old

Exclusion Criteria:

Receiving medical treatment for PMS Being pregnant or having experienced pregnancy before Having a systemic or chronic disease No physical or mental health problems that prevent exercise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female students over the age of 18
Enrollment: 72 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-07 (Estimated)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale | 10 weeks
  Premenstrual syndrome scale is a five-point Likert type scale consisting of 44 questions measuring the severity of premenstrual symptoms based on DSM-III and DSM-IV-R, in order to measure the severity of premenstrual symptoms by Gençdoğan (2006). In scoring the scale, the "Never" option is evaluated as 1 point, the "Very little" option as 2 points, the "Sometimes" option as 3 points, the "Often" option as 4 points, and the "Constantly" option as 5 points.
Depression Anxiety Stress Scale-21 | 10 weeks
  The DASS-21 scale, which is an abbreviated version of DASÖ-42 developed by Lovibond and Lovibond in 1995, was used. The 21-item short form (DASS-21) of the scale was adapted to Turkish by Sarıçam in 2018 in normal and clinical samples. The scale is a 4-point Likert-type scale and includes 21 questions in total, 7 questions each to measure the dimensions of depression, anxiety and stress.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Abiç, PhD, Principal Investigator — Eastern Mediterranean University; Sinem Dağ Canatan, MsC, Principal Investigator — Eastern Mediterranean University; Aslı Er Korucu, PhD, Principal Investigator — Ankara University; Ahu Aksoy Can, PhD, Principal Investigator — Mersin University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abic A, Dag-Canatan S, Er-Korucu A, Aksoy-Can A. The effects of yoga and progressive muscle relaxation exercises on premenstrual syndrome: a randomized controlled trial. Women Health. 2024 Mar;64(3):261-273. doi: 10.1080/03630242.2024.2314524. Epub 2024 Feb 11. PMID 38343144
- See also: Efficacy of a short-term yoga-based lifestyle intervention in reducing stress and inflammation: preliminary results. — http://pubmed.ncbi.nlm.nih.gov/22830969/
- See also: Effects of a Yoga Program on Menstrual Cramps and Menstrual Distress in Undergraduate Students with Primary Dysmenorrhea: A Single-Blind, Randomized Controlled Trial — http://pubmed.ncbi.nlm.nih.gov/27315239/